CLINICAL TRIAL: NCT00075465
Title: Phase II Study of Docetaxel and Epirubicine as First-Line Treatment in Patients With Advanced or Metastatic Adenocarcinoma of the Stomach
Brief Title: Docetaxel and Epirubicin as First-Line Therapy in Treating Patients With Locally Advanced or Metastatic Adenocarcinoma of the Stomach
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000346617; FRE-GERCOR-EPITAXD00-1; EU-20326
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2008-07-24 (Estimated); Status verified 2007-07

CONDITIONS: Gastric Cancer
Keywords: adenocarcinoma of the stomach; stage III gastric cancer; stage IV gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; Epirubicin

INTERVENTIONS:
Drug: docetaxel
Drug: epirubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and epirubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. Giving more than one drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving docetaxel together with epirubicin as first-line therapy works in treating patients with locally advanced or metastatic adenocarcinoma (cancer) of the stomach.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective tumor response rate and time to tumor progression in patients with locally advanced or metastatic adenocarcinoma of the stomach treated with docetaxel and epirubicin as first-line therapy.

Secondary

* Determine the survival without local relapse and overall survival of patients treated with this regimen.
* Determine the tolerance to this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive epirubicin IV over 30 minutes and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the stomach

  * Locally advanced or metastatic disease
* Measurable disease

  * At least 1 unidimensionally measurable target lesion at least 2 cm in diameter
* No known symptomatic brain metastases
* No bone metastases

PATIENT CHARACTERISTICS:

Age

* 18 to 75

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin less than 2 times normal
* AST and ALT no greater than 2.5 times normal
* Alkaline phosphatase no greater than 2.5 times normal

Renal

* Creatinine less than 1.6 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No serious cardiac failure within the past 12 months
* No myocardial infarction within the past 12 months
* No cardiac insufficiency
* No angina

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No uncontrolled serious infection
* No significant brain or psychiatric disorders
* No intolerance to cortisone or polysorbate 80
* No other prior malignancy except curatively treated basal cell skin cancer or carcinoma in situ of the cervix
* No other illness or medical condition that would preclude study participation
* No peripheral neuropathy greater than grade 2

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 21 days since prior participation in another clinical study
* No other concurrent experimental medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-04

PRIMARY OUTCOMES:
Objective tumor response rate
Time to tumor progression

SECONDARY OUTCOMES:
Survival without local relapse
Overall survival
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Louvet, MD, PhD — Hopital Saint Antoine
Locations (23):
- France (23):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospital General Robert Ballanger, Aulnay-sous-Bois
  - C.H.G. Beauvais, Beauvais
  - Clinique Tivoli, Bordeaux
  - Hopital Louis Pasteur, Chartres
  - Hopital Drevon, Dijon
  - Clinique Sainte-Marguerite, Hyères
  - Clinique Victor Hugo, Le Mans
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Clinique Saint Jean, Lyon
  - Hopital de la Croix Rousse, Lyon
  - CHU de la Timone, Marseille
  - Intercommunal Hospital, Montfermeil
  - American Hospital of Paris, Neuilly-sur-Seine
  - Hopital Saint Antoine, Paris
  - Hopital Saint Joseph, Paris
  - Hopital Tenon, Paris
  - Maison Medicale Marzet, Pau
  - Hopital Rene Dubos, Pontoise
  - C.H. Senlis, Senlis
  - Hopital d'Instruction des Armes Sainte-Anne, Toulon
  - CHRU de Tours - Hopital Trousseau, Tours